CLINICAL TRIAL: NCT02553421
Title: Optical Detection of Intravenous Infiltration:A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ivWatch, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IVW-CLR-CS09-400
Record Dates: First submitted 2015-09-16; First posted 2015-09-17 (Estimated); Results first posted 2017-01-05 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: Infiltration of Peripheral IV Therapy
Keywords: infiltration; extravasation; peripheral intravenous therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pilot (Experimental): A non-alarming ivWatch device will monitor the IV sites of these subjects. The goal of this small pilot study is to give clinicians an opportunity to perform the protocol and operate the ivWatch device and to give researchers the ability to make adjustments prior to starting the subsequent non-alarming group.
  Interventions: Device: ivWatch Model 400
- Non-alarming (Experimental): 150 patients will be enrolled in the non-alarming group. The ivWatch device will monitor the IV sites but will not issue infiltration notifications.
  Interventions: Device: ivWatch Model 400
- Alarming (Experimental): 150 patients will be enrolled in the alarming group. The IV sites will be monitored with the ivWatch Model 400 infiltration notifications enabled.
  Interventions: Device: ivWatch Model 400

INTERVENTIONS:
Device: ivWatch Model 400 — The ivWatch Model 400 is placed next to the subject's PIV site. All subjects will receive standard care for their IV sites including the normal routine assessments of the IV site by the bedside registered nurses.

SUMMARY:
This study will examine the use of the ivWatch Model 400 to monitor PIV sites in pediatric patients. Half the participants will be monitored by the device without infiltration notifications and the other half will be monitored by the device with infiltration notifications enabled.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent and/or assent
* Newborn to 17 years of age
* Weight > 2.5 kg

Exclusion Criteria:

* Severe skin integrity issues such as severe eczema, burns, epidermolysis bullosa, rash, hives
* Severe scarring of tissue (excessive IV use)
* Tattoo in area of PIV site
* IV site located in antecubital fossa

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 243 (Actual)
Dates: Start 2015-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-alarming: The ivWatch device will monitor the IV sites but will not issue infiltration notifications.
  ivWatch Model 400: The ivWatch Model 400 is placed next to the subject's PIV site. All subjects will receive standard care for their IV sites including the normal routine assessments of the IV site by the bedside registered nurses.
  Patients enrolled into the pilot and non-alarming portion of the study were combined for analysis due to no protocol changes between the study arms.
- Alarming: The IV sites will be monitored with the ivWatch Model 400 infiltration notifications enabled.
  ivWatch Model 400: The ivWatch Model 400 is placed next to the subject's PIV site. All subjects will receive standard care for their IV sites including the normal routine assessments of the IV site by the bedside registered nurses.
Period: Overall Study
Arm/Group | Non-alarming | Alarming
Started | 185 | 58
Completed | 156 | 57
Not Completed | 29 | 1
Not completed — Lost to Follow-up | 21 | 1
Not completed — Incomplete or Insufficient Data Collecte | 5 | 0
Not completed — Improper Device Placement | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-alarming | Alarming | Total
Number analyzed (Participants) | 185 | 58 | 243
Age, Continuous [Mean (Full Range); unit: years] | 7.61 [0.06 to 17] | 7.19 [0.04 to 17] | 7.51 [0.04 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 32 | 127
  Male | 90 | 26 | 116
IV Site [Number; unit: participants]
  Hand | 88 | 26 | 114
  Forearm | 81 | 32 | 113
  Leg/Foot | 12 | 0 | 12
  Other | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Time Infiltration Detected by Nurse
Description: The difference in time to detection between the clinician and the ivWatch device is measured from the non-alarming group. This measurement reveals how much earlier the infiltration could have been detected by the ivWatch device compared to the clinician assessments. This metric is measured using the patients in the non-alarming group since an infiltration notification by the ivWatch device could bias the clinician's diagnosis.
Time Frame: Participants will be followed for the duration of intravenous therapy, an expected duration of up to 1 week
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Non-alarming
Number analyzed (Participants) | 156
hours
  Red Notification | 29.8 [14.8 to 44.8]
  Yellow Notification | 32.3 [17.3 to 47.3]

2. Primary Outcome: Infiltration Sensitivity
Description: The infiltration sensitivity is defined as the percentage of the clinician-confirmed infiltrations that are detected by the ivWatch device before the clinician's diagnosis. This metric is measured and reported separately for non-alarming and alarming groups, since an infiltration notification by the ivWatch device could bias the clinician's diagnosis.
Time Frame: Participants will be followed for the duration of intravenous therapy, an expected duration of up to 1 week
Measure: Number (95% Confidence Interval); unit: percentage of infiltrations detected
Arm/Group | Non-alarming | Alarming
Number analyzed (Participants) | 156 | 57
percentage of infiltrations detected | 78.3 [56.5 to 92.5] | 80 [51.9 to 95.7]

3. Primary Outcome: Notification Rate of ivWatch Device
Description: The notification rate is defined as the number of ivWatch device infiltration notifications issued in a certain amount of time, typically reported in units of notifications per day. The notification rate is the number of notifications per day, excluding cases with clinician confirmed infiltrations. This metric is measured using the subjects in the alarming group since the number of notifications could potentially depend on how quickly nurses reset the device.
Time Frame: Participants will be followed for the duration of intravenous therapy, an expected duration of up to 1 week
Population: The number of participated in the Alarming group that did not have an infiltration diagnosed by a clinician.
Measure: Number (95% Confidence Interval); unit: Notifications per day
Arm/Group | Alarming
Number analyzed (Participants) | 42
Notifications per day
  Red Notifications | 0.280 [0.156 to 0.500]
  Yellow Notifications | 0.274 [0.119 to 0.631]

ADVERSE EVENTS:
Time Frame: Participants will be followed for the duration of intravenous therapy, an expected duration of up to 1 week
Arm/Group | Non-alarming | Alarming
Serious Adverse Events (participants affected / at risk) | 0/185 | 0/58
Other Adverse Events (participants affected / at risk) | 0/185 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less